CLINICAL TRIAL: NCT01019122
Title: Longitudinal Assessment of Bone Growth and Development in a Facility-Based Population of Children With Cerebral Palsy
Brief Title: Longitudinal Assessment of Bone Growth in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Collaborators: Kent State University (Other); University of North Carolina (Other); Alfred I. duPont Hospital for Children (Other)
Responsible Party: Richard Grossberg, MD, Hattie Larlham Center for Children with Disabilities
Other Study IDs: Bone Growth in CP Patients
Record Dates: First submitted 2009-11-20; First posted 2009-11-24 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Cerebral Palsy; Bone Density
Keywords: cerebral palsy; DEXA scan; bone density
MeSH Terms: conditions — Cerebral Palsy | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dexa Scan: Eligible patients from 2003 study will receive a follow-up Dexa scan.
  Interventions: Radiation: Dexa Scan

INTERVENTIONS:
Radiation: Dexa Scan — Dexa scan of left and right distal femur, then lumbar spine, and whole body when possible

SUMMARY:
In 2003, observational growth and bone density data was obtained on children with cerebral palsy (CP) living at Hattie Larlham as part of a study comparing growth with an existing database of children with CP who live at home. The original residents included in that study are now of adult age. Due to the lack of longitudinal bone density measurements in facility-based adults with severe CP, the investigators' objective is to obtain 6-year follow-up data from the residents enrolled in the original study.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Hattie Larlham Center for Children with Disabilities (HLCCD)
* Previously enrolled in the Growth in a Facility-Based Population of Children with Cerebral Palsy study in 2003

Exclusion Criteria:

* Resident of HLCCD who was not enrolled in the Growth in a Facility-Based Population of Children with Cerebral Palsy study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of a long-term care facility for children with disabilities who have severe to profound CP and are non-ambulatory.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Dual Energy X-ray Absorptiometry (DEXA) scan results | 6 years from original DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Martha Blackford, PharmD, Study Chair — Akron Children's Hospital; Michael Reed, PharmD, Study Chair — Akron Children's Hospital; Richard Henderson, MD, PhD, Study Chair — University of North Carolina